CLINICAL TRIAL: NCT01408498
Title: Study on the Effects of Exogenous Testosterone on Threat Perception and Behavioral Avoidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Scott Liening, Graduate Student, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SHL-Diss-1
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Testosterone's Effects on Threat Perception/Response
Keywords: Testosterone; Social psychology; Human behavior
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Control (No Intervention): Control group who will not receive exogenous testosterone administration. Will act as a comparison group to the testosterone group.
- Testosterone administration group (Experimental): Experimental group that will receive a single 10 g dose of 1% testosterone topical gel.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Topical administration of testosterone gel. Participants receive a one-time, single dose of 10 g of 1% testosterone gel.
  Other Names: AngroGel
  Arms: Testosterone administration group

SUMMARY:
The study aims to establish a clear causal link between testosterone and threat perception and behavioral responses to threat. Namely, the study focuses whether high levels of testosterone will cause an individual to exhibit increased physiological responses to threat (e.g., increased blood pressure, heart rate, and endocrine responses) and a decreased behavioral response (e.g., ignoring the threat, avoiding the threat, and postponing dealing with the threat). The threat in this study is a social threat involving public speaking, and is an outgrowth of previous research on the avoidance of health threats.

DETAILED DESCRIPTION:
Participants in the study will receive either a single dose of 10g 1% testosterone topical gel or placebo the day prior to participating in the study. The day of the study, participants will provide saliva samples throughout the study to track testosterone and cortisol levels. Participants will be asked to complete the Trier Social Stressor Task, which includes having to give a 5 minute speech to a panel of judges. Participants will be given the opportunity to postpone giving their speech to an unspecified date. The study will focus on two types of responses to the threat of public speaking: behavioral and physiological. The behavior of interest will be participants desire to postpone dealing with the threat (it is hypothesized that those in the testosterone administration group will have an increased desire to postpone). The physiological responses include increased levels of cortisol and increased cardiovascular tone (it is hypothesized that the testosterone administration group will show an increased physiological response compared to the placebo group).

ELIGIBILITY:
Inclusion Criteria:

* Male
* In good health
* Aged 18-35

Exclusion Criteria:

* Female
* Known carcinoma of the breast or prostate
* Known sensitivity to alcohol or soy products
* Preexisting cardiac, renal, or hepatic diseases
* Obesity
* Chronic lung diseases
* Cancer
* Use of anticoagulants
* Use of insulin or a history of diabetes
* Use of corticosteroids
* High levels of physical contact with women or children
* Preexisting liver problems

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Behavioral response | 16 hours post testosterone administration
  Participants will be asked to give a public speech, but will be given the opportunity to postpone the speech to a future date. Postponement is considered an avoidance-oriented behavioral response to a perceived social threat.
Physiological response | 16 hours post testosterone administration
  Participants will have cortisol and cardiovascular tone tracked during the social threat protocol. Prior to, during, and after being asked, preparing, and giving a public speech, participants' physiological stress markers will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Liening, B.A., Principal Investigator — University of Texas at Austin
Locations (1):
- Seay Building, Austin, Texas, United States